CLINICAL TRIAL: NCT04441255
Title: A Phase 1, Randomized, 2-Period, 2-Sequence, Crossover Study to Evaluate the Effect of High-Fat Meal on TAK-788 Pharmacokinetics in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of High-Fat Meal on TAK-788 Pharmacokinetics (PK) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-788-1005; CA24171 (Other: Celerion)
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-788 160 mg Fasted + TAK-788 160 mg Fed (Experimental): TAK-788 160 milligram (mg), capsule, orally, once on Day 1 of Period 1 under fasted conditions (Treatment A), followed by 10 days washout period, followed by TAK-788 160 mg, capsule, orally, once on Day 1 of Period 2 under fed conditions (Treatment B).
  Interventions: Drug: TAK-788
- TAK-788 160 mg Fed + TAK-788 160 mg Fasted (Experimental): TAK-788 160 mg, capsule, orally, once on Day 1 of Period 1 under fed conditions (Treatment B), followed by 10 days washout period, followed by TAK-788 160 mg, capsule, orally, once on Day 1 of Period 2 under fasted conditions (Treatment A).
  Interventions: Drug: TAK-788

INTERVENTIONS:
Drug: TAK-788 — TAK-788 Capsule.
  Other Names: AP32788; Mobocertinib

SUMMARY:
The purpose of this study is to characterize the effect of a high-fat meal on the PK of TAK-788 administered in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-788. The study will characterize the effect of a high-fat meal on the PK of TAK-788 administered in healthy participants.

The study will enroll approximately 14 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment sequence

* TAK-788 160 mg Fasted (Reference) in Period 1 + TAK-788 160 mg Fed (Test) in Period 2
* TAK-788 160 mg Fed (Test) in Period 1 + TAK-788 160 mg Fasted (Reference) in Period 2

All participants will be asked to take capsules of assigned TAK-788 on Day 1 of each period.

This single-center trial will be conducted in the United States. The overall time to participate in this study is 61 days. Participants will be contacted by telephone for 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non-smoker who has not used nicotine-containing products for at least 20 years prior to the first dosing and throughout the study, based on participant self-reporting.
2. Body mass index (BMI) greater than or equal to (>=) 18.5 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2), at screening.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiogram (ECGs), as deemed by the Investigator or designee.

Exclusion Criteria:

1. History of any illness (including hyperlipidemia and diabetes since high fat meal is required) that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
2. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
3. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
4. History or presence of any previous lung disease and/or current lung infection.
5. Positive urine drug or alcohol results at screening or first check-in.
6. Positive results at screening for Human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV).
7. Positive test result for active coronavirus disease 2019 (COVID-19).
8. Seated blood pressure is less than (<) 90/40 millimeter of mercury of mercury (mmHg) or greater than 140/90 mmHg at screening.
9. Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
10. QT interval corrected for heart rate using Fridericia's formula (QTcF) interval is greater than (>) 460 millisecond (msec) (males) or >470 msec (females) or ECG findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
11. Creatinine clearance <90 milliliter per minute (mL/min) at screening (calculated using the Cockcroft-Gault formula).
12. Unable to refrain from or anticipates the use of:

    o Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Medication listed as part of acceptable birth control methods will be allowed. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to the first dosing.

    Acetaminophen (up to 2 gram per 24 hour period) may be permitted during the study, only after initial dosing, if necessary, to treat adverse events (AEs).

    o Any drugs known to be inhibitors or inducers of Cytochrome P450 (CYP3A) enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, within 28 days prior to the first dosing and throughout the study.
13. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
14. Donation of blood or significant blood loss within 56 days prior to the first dosing.
15. Plasma donation within 7 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 01 July 2020 to 10 August 2020.
Pre-assignment Details: Healthy participants were enrolled in 1 of the 2 treatment sequences of this 2-period cross-over study to receive mobocertinib (TAK-788) 160 milligram (mg), capsule, in fasted condition (Treatment A) or mobocertinib 160 mg, capsule, in fed condition (Treatment B).
Groups:
- Mobocertinib 160 mg Fasted + Mobocertinib 160 mg Fed: Mobocertinib 160 mg, capsule, orally, once on Day 1 of Period 1 under fasted conditions (Treatment A), followed by 10 days washout period, further followed by mobocertinib 160 mg, capsule, orally, once on Day 1 of Period 2 under fed conditions (Treatment B).
- Mobocertinib 160 mg Fed + Mobocertinib 160 mg Fasted: Mobocertinib 160 mg, capsule, orally, once on Day 1 of Period 1 under fed conditions (Treatment B), followed by 10 days washout period, further followed by mobocertinib 160 mg, capsule, orally, once on Day 1 of Period 2 under fasted conditions (Treatment A).
Period: Period 1 (1 Day)
Arm/Group | Mobocertinib 160 mg Fasted + Mobocertinib 160 mg Fed | Mobocertinib 160 mg Fed + Mobocertinib 160 mg Fasted
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout Period (10 Days)
Arm/Group | Mobocertinib 160 mg Fasted + Mobocertinib 160 mg Fed | Mobocertinib 160 mg Fed + Mobocertinib 160 mg Fasted
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Period 2 (1 Day)
Arm/Group | Mobocertinib 160 mg Fasted + Mobocertinib 160 mg Fed | Mobocertinib 160 mg Fed + Mobocertinib 160 mg Fasted
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least one dose of a study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobocertinib 160 mg Fasted + Mobocertinib 160 mg Fed | Mobocertinib 160 mg Fed + Mobocertinib 160 mg Fasted | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (9.61) | 35.4 (9.14) | 34.7 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 73.89 (11.879) | 76.70 (16.416) | 75.29 (13.843)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 174.3 (9.48) | 175.6 (13.50) | 174.9 (11.23)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.293 (3.0143) | 24.706 (3.2743) | 24.499 (3.0311)

OUTCOME MEASURES:

1. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Median (Full Range); unit: hours
Groups:
- Mobocertinib 160 mg Fasted: Mobocertinib 160 mg, capsule, orally, once on Day 1 of either Period 1 or Period 2 under fasted conditions (Treatment A).
- Mobocertinib 160 mg Fed: Mobocertinib 160 mg, capsule, orally, once on Day 1 of either Period 1 or Period 2 under fed conditions (Treatment B).
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
hours | 6.01 [4.00 to 8.00] | 8.00 [4.01 to 12.0]

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
nanogram per milliliter (ng/mL) | 56.8 (47.1) | 56.6 (40.9)

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
nanogram*hour per milliliter (ng*hr/mL) | 1030 (61.1) | 1230 (59.5)

4. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
ng*hr/mL | 1020 (61.4) | 1210 (60.0)

5. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Active Metabolites (AP32960 and AP32914) of Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Median (Full Range); unit: hours
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
hours
  AP32960 | 6.00 [4.00 to 8.02] | 8.00 [4.01 to 8.08]
  AP32914 | 6.01 [4.00 to 8.02] | 8.00 [4.01 to 12.1]

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Active Metabolites (AP32960 and AP32914) of Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
ng/mL
  AP32960 | 31.1 (22.3) | 27.7 (22.5)
  AP32914 | 4.34 (31.7) | 3.73 (31.8)

7. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Active Metabolites (AP32960 and AP32914) of Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Here "number analyzed" were participants who were evaluable for the outcome measure at given categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
ng*hr/mL
  AP32960 | 704 (31.3) | 731 (32.2)
  AP32914: number analyzed (Participants) | 12 | 11
  AP32914 | 79.4 (47.4) | 89.2 (50.6)

8. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Active Metabolites (AP32960 and AP32914) of Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: The PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
Number analyzed (Participants) | 13 | 14
ng*hr/mL
  AP32960 | 682 (31.9) | 709 (32.7)
  AP32914 | 69.2 (50.1) | 72.2 (53.9)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug until 30 days after last dose of study drug in Period 2 (up to Day 42).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Mobocertinib 160 mg Fasted | Mobocertinib 160 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobocertinib 160 mg Fasted (N=14) | Mobocertinib 160 mg Fed (N=14)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Feeling abnormal (General disorders) | 0 | 1
Feeling cold (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Pustule (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04441255/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04441255/SAP_001.pdf